CLINICAL TRIAL: NCT03878524
Title: Serial Measurements of Molecular and Architectural Responses to Therapy (SMMART) Trial: PRIME
Brief Title: Serial Measurements of Molecular and Architectural Responses to Therapy (SMMART) PRIME Trial
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lara Davis, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015588; NCI-2020-02743 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00015588 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Anatomic Stage IV Breast Cancer AJCC v8; Anemia; Ann Arbor Stage III Hodgkin Lymphoma; Ann Arbor Stage III Non-Hodgkin Lymphoma; Ann Arbor Stage IV Hodgkin Lymphoma; Ann Arbor Stage IV Non-Hodgkin Lymphoma; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Castration-Resistant Prostate Carcinoma; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphoid System Neoplasm; Locally Advanced Pancreatic Adenocarcinoma; Metastatic Breast Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Pancreatic Adenocarcinoma; Myelodysplastic/Myeloproliferative Neoplasm With Ring Sideroblasts and Thrombocytosis; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Primary Myelofibrosis; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Hematologic Malignancy; Recurrent Hodgkin Lymphoma; Recurrent Myelodysplastic Syndrome; Recurrent Myelodysplastic/Myeloproliferative Neoplasm; Recurrent Myeloproliferative Neoplasm; Recurrent Non-Hodgkin Lymphoma; Recurrent Plasma Cell Myeloma; Recurrent Small Lymphocytic Lymphoma; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Chronic Myelomonocytic Leukemia; Refractory Hematologic Malignancy; Refractory Hodgkin Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Myelodysplastic Syndrome; Refractory Myelodysplastic/Myeloproliferative Neoplasm; Refractory Non-Hodgkin Lymphoma; Refractory Plasma Cell Myeloma; Refractory Primary Myelofibrosis; Refractory Small Lymphocytic Lymphoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Unresectable Pancreatic Adenocarcinoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Anemia; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Breast Neoplasms; Neoplasm Metastasis; Thrombocytosis; Myeloproliferative Disorders; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hematologic Neoplasms; Hodgkin Disease; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Myelomonocytic, Chronic; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — abemaciclib; abiraterone; Afatinib; Bevacizumab; Immunoglobulin G; Disulfides; bicalutamide; Specimen Handling; Bortezomib; cabazitaxel; XRP6258; cabozantinib; Capecitabine; Carboplatin; Celecoxib; cobimetinib; copanlisib; dabrafenib; dacomitinib; darolutamide; Dasatinib; Doxorubicin; durvalumab; enasidenib; entrectinib; enzalutamide; Erlotinib Hydrochloride; Everolimus; Fluorouracil; dehydroftorafur; idelalisib; Imatinib Mesylate; Ipilimumab; CTLA-4 Antigen; lenvatinib; Leucovorin; lorlatinib; Losartan; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; neratinib; Nivolumab; olaparib; Oxaliplatin; palbociclib; Panobinostat; pembrolizumab; pertuzumab; 2C4 antibody; ponatinib; regorafenib; ruxolitinib; Sirolimus; Sorafenib; Sunitinib; trametinib; Ado-Trastuzumab Emtansine; Tretinoin; Vemurafenib; venetoclax; HhAntag691; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (biospecimen collection, 2 drug combination) (Experimental): TUMOR BIOPSY: Patients undergo collection of tissue samples. Clinical analytics are performed on the samples and analyzed by a clinical tumor board to recommend a treatment option based on those analytics.
  SMMART-PRIME TREATMENT: Patients receive a combination of 2 drugs (Drug A and Drug B, selected from interventions below). Doses will be escalated within individual patients over time. As described in detail below, escalation will occur monthly and is anticipated to occur as follows: first month - 100% FDA approved dose Drug A + 25% FDA approved dose Drug B; second month -- 100% dose Drug A + 50% dose Drug B; third month -- 100% dose Drug A + 100% dose Drug B. All dose-escalations will be reviewed and approved by an independent consultant outside of Oregon Health & Science University (OHSU).
  Treatment will continue for up to the end of 6 treatment cycles (cycle length is between 21-28 days) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Drug: Abiraterone; Drug: Afatinib; Biological: Bevacizumab; Drug: Bicalutamide; Procedure: Biospecimen Collection; Drug: Bortezomib; Drug: Cabazitaxel; Drug: Cabozantinib; Drug: Capecitabine; Drug: Carboplatin; Drug: Celecoxib; Drug: Cobimetinib; Drug: Copanlisib; Drug: Dabrafenib; Drug: Dacomitinib; Drug: Darolutamide; Drug: Dasatinib; Drug: Doxorubicin; Biological: Durvalumab; Drug: Enasidenib; Drug: Entrectinib; Drug: Enzalutamide; Drug: Erlotinib; Drug: Everolimus; Drug: Fluorouracil; Drug: Idelalisib; Drug: Imatinib; Biological: Ipilimumab; Drug: Lenvatinib; Drug: Leucovorin; Drug: Lorlatinib; Drug: Losartan; Drug: Nab-paclitaxel; Drug: Neratinib; Biological: Nivolumab; Drug: Olaparib; Drug: Oxaliplatin; Drug: Palbociclib; Drug: Panobinostat; Biological: Pembrolizumab; Biological: Pertuzumab; Drug: Ponatinib; Other: Quality-of-Life Assessment; Drug: Regorafenib; Drug: Ruxolitinib; Drug: Sirolimus; Drug: Sorafenib; Drug: Sunitinib; Drug: Trametinib; Biological: Trastuzumab Emtansine; Drug: Tretinoin; Drug: Vemurafenib; Drug: Venetoclax; Drug: Vismodegib; Drug: Vorinostat

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
Drug: Abiraterone — Given PO
  Other Names: CB 7598
Drug: Afatinib — Given PO
  Other Names: BIBW 2992; BIBW2992
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev; Anti-VEGF Monoclonal Antibody SIBP04; SIBP 04; SIBP-04; SIBP04
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Procedure: Biospecimen Collection — Undergo collection of biospecimens (including tissue, blood, or previously collected archival specimens)
  Other Names: Biological Sample Collection; Specimen Collection
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Cabazitaxel — Given IV
  Other Names: Jevtana; RPR-116258A; Taxoid XRP6258; XRP-6258
Drug: Cabozantinib — Given PO
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Celecoxib — Given PO
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; SC-58635; YM 177
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518; 934660-93-2
Drug: Copanlisib — Given IV
  Other Names: BAY 80-6946; PI3K Inhibitor BAY 80-6946
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436; GSK-2118436A; GSK2118436
Drug: Dacomitinib — Given PO
  Other Names: EGFR Inhibitor PF-00299804; PF-00299804; PF-00299804-03; PF-299804; Vizimpro
Drug: Darolutamide — Given PO
  Other Names: Antiandrogen ODM-201; BAY 1841788; BAY-1841788; BAY1841788; Nubeqa; ODM 201; ODM-201; 1297538-32-9
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736; 1428935-60-7
Drug: Enasidenib — Given PO
  Other Names: AG-221; CC-90007 Free Base
Drug: Entrectinib — Given PO
  Other Names: Rozlytrek; RXDX 101; RXDX-101; RXDX101
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Drug: Erlotinib — Given PO
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Idelalisib — Given PO
  Other Names: CAL-101; GS 1101; GS-1101; Phosphoinositide-3 Kinase Delta Inhibitor CAL-101; Zydelig
Drug: Imatinib — Given PO
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Drug: Lenvatinib — Given PO
  Other Names: E7080; ER-203492-00; Multi-Kinase Inhibitor E7080
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Lorlatinib — Given PO
  Other Names: 2H-4,8-Methenopyrazolo(4,3-H)(2,5,11)benzoxadiazacyclotetradecine-3-carbonitrile, 7-amino-12-fluoro-10,15,16,17-tetrahydro-2,10,16-trimethyl-15-oxo-, (10R)-; Lorbrena; PF-06463922
Drug: Losartan — Given PO
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
Drug: Neratinib — Given PO
  Other Names: (2E)-N-(4-((3-chloro-4-((pyridin-2-yl)methoxy)phenyl)amino)-3-cyano-7-ethoxyquinolin-6-yl)-4-(dimethylamino)but-2-enamide; HKI 272; HKI-272; PB 272; PB-272
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991
Drug: Panobinostat — Given PO
  Other Names: Faridak; LBH589
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar HS627; rhuMAb2C4; RO4368451; HLX11
Drug: Ponatinib — Given PO
  Other Names: AP-24534; AP24534
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; REGORAFENIB ANHYDROUS; Stivarga
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Jakafi; Oral JAK Inhibitor INCB18424
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217
Drug: Sorafenib — Given PO
  Other Names: BA4 43 9006; BAY 43-9006; Bay-439006
Drug: Sunitinib — Given PO
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212
Biological: Trastuzumab Emtansine — Given IV
  Other Names: Ado Trastuzumab Emtansine; ADO-Trastuzumab Emtansine; Kadcyla; PRO132365; RO5304020; T-DM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate
Drug: Tretinoin — Given PO
  Other Names: 2,4,6,8-Nonatetraenoic acid, 3, 7-dimethyl-9-(2,6,6-trimethyl-1-cyclohexen-1-yl)-, (all-E)-; Aberel; Airol; Aknoten; all trans-Retinoic acid; All-trans Retinoic Acid; All-trans Vitamin A Acid; all-trans-Retinoic acid; all-trans-Vitamin A acid; ATRA; Avita; beta-Retinoic Acid; Cordes Vas; Dermairol; Epi-Aberel; Eudyna; Renova; Retin-A; Retin-A MICRO; Retin-A-Micro; Retinoic Acid; Retisol-A; Ro 5488; Stieva-A; Stieva-A Forte; Trans Retinoic Acid; Trans Vitamin A Acid; trans-Retinoic Acid; Tretinoinum; Vesanoid; Vitamin A Acid; Vitamin A acid, all-trans-; Vitinoin
Drug: Vemurafenib — Given PO
  Other Names: BRAF (V600E) kinase inhibitor RO5185426; BRAF(V600E) Kinase Inhibitor RO5185426; PLX-4032; PLX4032; RG 7204; RG7204; RO 5185426; Zelboraf
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase Ib trial determines if samples from a patient's cancer can be tested to find combinations of drugs that provide clinical benefit for the kind of cancer the patient has. This study is also being done to understand why cancer drugs can stop working and how different cancers in different people respond to different types of therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of implementing an individualized treatment strategy for advanced solid tumor and hematological malignancies based upon a comprehensive assessment of tumor and patient characteristics.

SECONDARY OBJECTIVES:

I. To describe the tolerability of implementing an individualized treatment strategy, particularly by measuring unanticipated toxicity associated with the administration of different combinations of two therapeutic agents given to an individual participant.

II. To assess the duration of treatment for participants receiving Serial Measurements of Molecular and Architectural Responses to Therapy (SMMART)-PRIME Therapy #1.

III. To determine overall survival of participants with advanced solid tumors and hematological malignancies.

IV. To determine the time to decline in a participant's ability to perform activities of daily living.

EXPLORATORY OBJECTIVES:

I. To measure quality of life among enrolled participants. II. To evaluate immune-mediated tumor response among participants receiving an immunomodulatory study drug.

III. To determine the rates of response and benefit to SMMART-PRIME Therapy #1, as an individualized treatment strategy for participants with advanced solid tumor and hematological malignancies.

IV. To determine the progression-free and disease-free survival of participants with advanced solid tumors and hematological malignancies.

OUTLINE:

TUMOR BIOPSY: Patients undergo collection of tissue samples. Clinical analytics are performed on the samples and analyzed by a clinical tumor board to recommend a treatment option based on those analytics. The findings from these Clinical Study Analytics are intended to provide the basis for selection of two drugs that, when administered in combination, provide an optimal and individualized treatment approach. This may or may not include a SMMART-PRIME treatment. The decision to initiate any SMMART-PRIME Therapy ultimately resides with the treating physician in conjunction with the study participant.

SMMART-PRIME TREATMENT: Patients receive a combination of 2 drugs (Drug A and Drug B, selected from interventions below). Doses will be escalated within individual patients over time. As described in detail below, escalation will occur on a monthly basis and is anticipated to occur as follows: first month -- 100% Food and Drug Administration (FDA) approved dose Drug A + 25% FDA approved dose Drug B; second month -- 100% dose Drug A + 50% dose Drug B; third month -- 100% dose Drug A + 100% dose Drug B. All dose-escalations will be reviewed and approved by an independent consultant outside of Oregon Health & Science University (OHSU).

Treatment will continue for up to the end of 6 treatment cycles (cycle length is between 21-28 days) in the absence of disease progression or unacceptable toxicity. Patients whose treatment is discontinued as a result of excess toxicity or lack of efficacy may switch to a different combination of drugs. Beyond six cycles, participants will be considered off-protocol directed treatment, and will move into long term follow-up.

After completion of study treatment, patients are followed for up to 5 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Participants >= 21 years old at time of informed consent. Both men and women and members of all races and ethnic groups will be included
* Participants, both men and women, must agree to use an adequate method of contraception prior to study entry, for the duration of study participation, and for 4 months after completion of study
* Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to start of study drug administration
* Patients must have a histologically or cytologically-confirmed metastatic solid tumor or hematological malignancy that has progressed as follows:

  * Patients with a solid tumor must have metastatic disease and have progressed on at least 1 line of established therapy that is known to provide clinical benefit, or for whom no standard curative therapy exists. Participants with newly diagnosed, unresectable, locally-advanced or metastatic pancreatic adenocarcinoma and are beginning first-line treatment with a course of chemotherapy are eligible OR
  * Participants must have a hematological malignancy that is advanced, relapsed, or refractory to at least 1 line of established therapy that is known to provide clinical for the treatment of their disease. Hematological disease included in this study are as follows:

    * Acute myelogenous leukemia (AML), or
    * Myelodysplastic syndrome (MDS), or
    * MDS/myeloproliferative neoplasms (MDS/MPN), or
    * Primary myelofibrosis (PMF)
    * Acute lymphoblastic leukemia (ALL)
    * Chronic myelogenous leukemia (CML)
    * Non-Hodgkin lymphoma (NHL) or Hodgkin's disease (HD)
    * Chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL)
    * Multiple myeloma (MM)
* Participants with a metastatic solid tumor or advanced hematological malignancy whom, due to medical issues cannot receive standard therapy shown to prolong survival, will be eligible, if other eligibility criteria are met

  * Patients with a metastatic solid tumor or advanced hematological malignancy that actively refuse chemotherapy that is considered standard treatment for their cancer, despite being informed by the investigator about the treatment options, are eligible for this study on a case-by-case basis (in consultation with the principal investigator [PI]). Potential participants actively refusing chemotherapy must have had progression or refractory disease prior to starting study treatment, and their refusal must be documented
* Participants must have measurable disease:

  * Patients with solid tumors must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. At least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, per RECIST (v1.1)
  * Note: Participants with lesions on a bone scan that are considered distinctly metastatic will also be included
  * Patients with lymphoma must have at least one non-irradiated tumor mass > 15 mm (long axis of lymph node) or > 10 mm (short axis of lymph node or extranodal lesions) on spiral CT-scan
  * Patients with CLL must have presence of radiographically measurable lymphadenopathy (defined as the presence of >= 1 nodal lesion that measures >= 2.0 cm in the longest diameter [LD] and >= 1.0 cm in the longest perpendicular diameter [LPD] as assessed by CT or magnetic resonance imaging [MRI])
  * Patients with MM must have at least one of the following: serum monoclonal component > 1 g/dL (IgG), or > 0.5 g/dL (IgA), or Bence-Jones (BJ) proteinuria > 200 mg/24 hour, or measurable plasmacytoma (not previously irradiated)
* Participants with a hematological malignancy must have their bone marrow biopsy and aspirate reviewed at Oregon Health & Science University (OHSU)
* Participants with a solid tumor must have lesions meeting the above criteria also and must be amenable to biopsy procedures performed per institutional standards
* Participants must not currently be receiving any other investigational agents
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2 and a physician assessed life expectancy of >= 6 months
* Absolute neutrophil count (ANC) >= 1,500/mcL (at time of registration and within 4 weeks prior to initiating on-protocol treatment)

  * Waived for those with hematological malignancy; and may be waived on a case-by-case basis for patient populations recognized to have normal baseline values below this level
* Platelets >= 100,000/mcL (at time of registration and within 4 weeks prior to initiating on-protocol treatment)

  * Waived for those with hematological malignancy
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (at time of registration and within 4 weeks prior to initiating on-protocol treatment)

  * Waived for those with hematological malignancy
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min/1.73 m^2 for participants with creatinine levels > 1 x institutional ULN (at time of registration and within 4 weeks prior to initiating on-protocol treatment)

  * Waived for those with hematological malignancy; and may be waived on a case-by-case basis for patient populations recognized to have normal baseline values below this level
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (at time of registration and within 4 weeks prior to initiating on-protocol treatment)

  * Creatinine clearance should be calculated per institutional standard. For participants with a baseline calculated creatinine clearance below normal institutional laboratory values, a measured baseline creatinine clearance should be determined. Individuals with higher values felt to be consistent with inborn errors of metabolism will be considered on a case-by-case basis
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (at time of registration and within 4 weeks prior to initiating on-protocol treatment)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (at time of registration and within 4 weeks prior to initiating on-protocol treatment)
* Activated partial thromboplastin time (aPTT) or PTT =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (at time of registration and within 4 weeks prior to initiating on-protocol treatment)
* Body mass index (BMI) > > 16.0 and < 35.0 kg/m^2 (at time of registration and within 4 weeks prior to initiating on-protocol treatment)

  * Participants with a BMI of >= 30.0 will use ideal body weight indices in calculating the delivery of agents that are dosed based upon body surface area (i.e., mg agent/meter squared) or weight (i.e., mg agent/kg body weight)
* Any prior therapy, radiotherapy (except palliative radiation therapy of 30 Gy or less), or major surgery must have been completed >= 4 weeks prior to start of study treatment. All adverse events due to prior therapy must have resolved to a grade 1 or better (except alopecia and lymphopenia for all disease cohorts, and hematologic toxicity for those with a hematological malignancy) by start of treatment. Palliative radiation therapy must have been completed at least 2 weeks prior to start of treatment. The radiotherapy must not be to a lesion that is included as measurable disease
* Additional cancer-specific inclusion criteria must also be met

Key Exclusion Criteria:

* Participants with metastases to the central nervous system that are considered uncontrolled and/or were diagnosed within the past 4 weeks of screening for this study
* Participants cannot have an active malignancy of another cancer. Those with a history of prior malignancy will be considered on a case-by-case basis. Guiding examples for those who can be enrolled include: individuals who have been disease free for > 5 years; individuals who are considered to have a high likelihood of being cured (e.g., prior history of stage 1 rectal cancer and currently otherwise disease free); adequately treated localized non-melanomatous skin cancer
* Participants cannot be on other forms of anti-cancer therapy at the same time, except as described within this protocol. There must be at least a washout period that accounts for 5 half-lives (or >= 21 days, whichever is longer) of last therapy

  * Participants with prostate cancer (PCa) will continue treatment with androgen deprivation therapy, either by prior castration or treatment with luteinizing hormone-releasing hormone (LHRH) antagonists or agonists, as is standard practice
  * Participants with breast cancer (BCa) who are HER2 positive may continue to receive anti-HER2 therapy per standard practice guidelines, while participants who are hormone receptor positive may continue to receive hormone therapy per standard practice guidelines
  * Participants with a hematological malignancy may continue to receive hydroxyurea or other hypomethylating agent for two cycles of SMMART-PRIME therapy, as described in this protocol
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure
* Chronic graft versus host disease (GVHD) or on immunosuppressive therapy for the control of GVHD
* Participants with uncontrolled infection will not be enrolled until infection is treated
* Participant is seropositive with human immunodeficiency virus (HIV) or has active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
  * For patients with evidence of chronic HBV infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
  * Individuals with a history of HCV infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Participants with medical conditions, inclusive of psychiatric, that in the opinion of the investigators would jeopardize the patient or the study will be excluded
* Participants that are pregnant or breast feeding
* ON-TREATMENT: Individuals that have medical and/or psychiatric conditions that in the opinion of investigators would jeopardize participant safety or study integrity if they were to receive on-study treatment will not proceed further treatment and will be removed from study
* ON-TREATMENT: If performance status is ECOG > 2
* ON-TREATMENT: History of allergic reaction to a recommended study agent or its excipients
* Additional cancer-specific exclusion criteria requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing an individualized treatment strategy (number of participants to receive first dose) | From date of tumor board recommendation to first dose of SMMART-PRIME Therapy #1 (up to 3 months)
  Measured as the number of participants to receive the first dose of Serial Measurements of Molecular and Architectural Responses to Therapy (SMMART)-PRIME therapy (Therapy #1) within 3 months from the date of Clinical Tumor Board providing a recommended drug combination.

SECONDARY OUTCOMES:
Incidence of grade 3+ toxicities attributable to assigned study drug(s) | 30 days post completion of each SMMART-PRIME Therapy (up to 6 months)
  Measured with National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Criteria version 5.0.
Time to treatment discontinuation | Completion of SMMART-PRIME Therapy #1 (up to 6 months)
  Measured as time (days) from start of SMMART-PRIME Therapy #1 to discontinuation for any reason.
Overall survival (OS) | Death from any cause (up to 60 months after the last dose of SMMART-PRIME Therapy #1)
  Overall survival (OS) is defined as the time (days) from start of SMMART-PRIME Therapy #1 to death from any reason.
Time to decline (TTD) | Completion of SMMART-PRIME Therapy #1 (up to 6 months)
  Measured time (days) from start of SMMART-PRIME Therapy #1 to recorded Eastern Cooperative Oncology Group (ECOG) performance status >= 3 using cumulative incidence methods.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Davis, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States